CLINICAL TRIAL: NCT01058772
Title: GINEXMAL RCT: Induction of Labour Versus Expectant Management in Gestational Diabetes Pregnancies
Brief Title: Gestational Diabetes: Induction Versus Expectant Management of Labour
Acronym: GINEXMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, Dr, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RC 22/09
Record Dates: First submitted 2010-01-26; First posted 2010-01-29 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Gestational Diabetes; Gestational Diabetes Mellitus; Diabetes Mellitus, Gestational; Pregnancy-Induced Diabetes; Diabetes, Pregnancy Induced
Keywords: Induced Labour; Expectant Management; C-section rate; Maternal Outcomes; Neonatal Outcomes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Labor, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INDUCTION of LABOUR (Experimental): At enrollment patients assigned to the induction group will be admitted to the obstetric ward and will undergo induction of labour as described in the intervention section.
  Once patient's Bishop score exceeds 7 or regular contractions are diagnosed, patients will be transferred to the delivery ward for artificial rupture of membranes (ARM) or Oxytocin augmentation as indicated.
  Interventions: Other: INDUCTION of LABOUR
- EXPECTANT MANAGEMENT (No Intervention): Patients enrolled in the conservative management arm will be followed up twice weekly for foetal wellbeing by Non-stress test and Biophysical profile. Patients will be followed up to 41+0 weeks.
  Patients, who will not deliver by this gestational age, will be admitted for labour induction (see the above protocol). Induction of labour will be offered when non-reassuring foetal status is suspected. All patients in the conservative arm will undergo foetal weight ultrasound estimation prior to induction. Patients with estimated foetal weight over 4000 gr will be offered a C-section.

INTERVENTIONS:
Other: INDUCTION of LABOUR — Induction of labour will be performed by using dinoprostone 2 mg vaginally or dinoprostone 0.5 mg intracervically at 6-8h interval (up to 5 doses) or dinoprostone 10 mg vaginal device. Patients, in which cervical ripening does not occur (Bishop score < 7) after 5 attempts with PGE2, will be offered either oxytocin or Foley catheter induction or C-section, according to local protocols.
  Arms: INDUCTION of LABOUR

SUMMARY:
The purpose of this study is to determine whether, in Gestational Diabetes Mellitus (GDM) pregnancies, induction of labour at 38-39 weeks of pregnancy is superior to expectant management in terms of maternal and neonatal outcomes.

DETAILED DESCRIPTION:
Gestational Diabetes Mellitus (GDM) is one of the most common complications of pregnancy and its incidence is estimated as around 7%. Babies born from women with GDM are significantly more exposed to perinatal risk. Furthermore in GDM pregnancies an increased C-section rate has been observed, mostly unjustified.

Strong evidence, based on prospective studies and randomized controlled trials, in favour or against the effectiveness and safeness of induction in women with GDM, are missing. The aim of the present study is to identify the best management for these women at term and provide evidence that could change the current clinical practice.

To reach this objective, 1760 eligible women will be recruited at 9 Teaching Hospitals (5 in Italy, 4 all over the world). Sample size has been estimated to demonstrate a difference between the two arms ≥ 6% (31% of C-section in the expectant group and 25% in the induction group; relative difference between the 2 groups equal to 20% in favor of induction; Kjos et al, 1993), considering an α error equal to 5% and 80% power.

Patients will be randomized to induction of labour (N=880) or expectant management (N=880). Data on maternal and neonatal outcomes will be collected at delivery and until maternal and neonatal discharge.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > 18;
* Singleton pregnancy in vertex presentation;
* Gestational age between 38-39 weeks verified by LMP and first trimester ultrasound when available;
* Women diagnosed with GDM in the current pregnancy [Diagnosis will be based upon abnormal 50 Gr. GCT (>140) followed by >2 abnormal indices in the OGTT (according to C&C criteria). Women with GCT>200 mg/dl will undergo 100 gr OGTT as well];
* No other contraindications for vaginal delivery.

Exclusion Criteria:

* Pre-gestational diabetes;
* Prior C-section;
* Suspected estimated fetal weight> 4000 gr. at enrollment;
* Any known contraindications for vaginal delivery;
* Uncertain gestational age;
* Non-reassuring fetal status necessitating immediate obstetrical intervention (prompt delivery/prompt C-section);
* Maternal disease complicating pregnancy and necessitating delivery (e.g Severe PET);
* Bishop score >7 at enrollment;
* Major fetal malformation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
C-section rate | 1 minute after delivery

SECONDARY OUTCOMES:
Operative Vaginal Delivery | 1 minute after delivery
Perineal Tears or Episiotomy | 1 minute after delivery
Postpartum haemorrhage | within 24 hours from delivery
Maternal Blood Transfusion | until maternal discharge
Maternal Intensive Care Unit Admission | until maternal discharge
Neonatal Weight | 10 minutes after delivery
Neonatal Apgar score at 1', 5', 10' minutes | 1, 5, 10 minutes after delivery
Shoulder Dystocia | during delivery
Manoeuvres for Shoulder Dystocia | during delivery
Neonatal Intensive Care Unit Admission | until neonatal discharge
Arterial cord Ph inferior to 7.2 | within 5 minutes from delivery
Neonatal Hyperbilirubinemia | until neonatal discharge
Clinical and Biochemical Neonatal Hypoglycemia | until neonatal discharge
Neonatal Polycythemia | until neonatal discharge
Neonatal Birth Trauma | 10 minute from delivery or until neonatal discharge
Neonatal Respiratory Distress/Transient Tachypnea | until neonatal discharge
Neonatal Need for Respiratory Support | until neonatal discharge
Maternal death | until neonatal discharge
Perinatal Death | until neonatal discharge
Spontaneous/Instrumental third stage of labour | within 1 hours from delivery
Indication for Cesarean Section | 1 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Alberico, MD, Study Director — Institute for Maternal and Child Health IRCCS Burlo Garofolo; Moshe Hod, MD, Study Director — Helen Schneider's Hospital for Women - Rabin Medical Center
Locations (9):
- Helen Schneider's Hospital for Women - Rabin Medical Center, Petah Tikva, Israel
- Italy (5):
  - I Ostetricia Spedali Civili, Brescia
  - Department of Gynecology Perinatology and Human Reproduction, Florence
  - Unità Operativa di Ostetricia e Ginecologia - Ospedale Buzzi, Milan
  - Institute for Maternal and Child Health - IRCCS Burlo Garofolo, Trieste
  - Dipartimento di Discipline Ginecologiche ed Ostetriche - Università di Torino, Turin
- Division Woman and Baby - UMC Utrecht/ Wilhelmina Children's Hospital, Utrecht, Netherlands
- Department of ob/gyn, Division of perinatology - University Medical Centre, Ljubljana, Slovenia
- Department of Obstetrics and Gynecology - University of Colombo, Colombo, Sri Lanka

REFERENCES:
- [Background] Maso G, Alberico S, Wiesenfeld U, Ronfani L, Erenbourg A, Hadar E, Yogev Y, Hod M; GINEXMAL Study Cooperative Research Group. "GINEXMAL RCT: Induction of labour versus expectant management in gestational diabetes pregnancies". BMC Pregnancy Childbirth. 2011 Apr 20;11:31. doi: 10.1186/1471-2393-11-31. PMID 21507262